CLINICAL TRIAL: NCT01646281
Title: Effects of Vernakalant and Flecainide on Atrial Contractility in Patients With Atrial Fibrillation
Brief Title: Vernakalant Versus Flecainide: Atrial Contractility
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL39854.068.12
Record Dates: First submitted 2012-07-09; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Vernakalant; Flecainide; Echocardiography
MeSH Terms: conditions — Atrial Fibrillation | interventions — vernakalant; Flecainide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flecainide (Active Comparator): Patients randomized to flecainide will receive a 10-minute infusion of 2 mg/kg (maximal 150 mg) flecainide. If the patient is still in AF 1 hour after the infusion, electrical cardioversion will be performed according to protocol.
  Interventions: Drug: Flecainide
- Vernakalant (Active Comparator): Patients randomized to vernakalant will receive a 10-minute infusion of 3 mg/kg vernakalant, followed by a 15 minute observation period. If the patient is still in atrial fibrillation, an additional 10-minute infusion of 2 mg/kg vernakalant will be given. If the patient is still in AF 1 hour after the infusion, electrical cardioversion will be performed according to protocol.
  Interventions: Drug: Vernakalant

INTERVENTIONS:
Drug: Vernakalant — 10-minute infusion of 3 mg/kg vernakalant, followed by a 15 minute observation period. If the patient is still in atrial fibrillation, an additional 10-minute infusion of 2 mg/kg vernakalant will be given.
  Other Names: Brinavess, EV product code SUB30707
  Arms: Vernakalant
Drug: Flecainide — 10-minute infusion of 2 mg/kg (maximal 150 mg)
  Other Names: Tambocor, EV product code SUB13894MIG
  Arms: Flecainide

SUMMARY:
Atrial fibrillation (AF) is associated with decreased atrial contractility which is associated with stroke. Decreased contractility becomes apparent after cardioversion of atrial fibrillation, a short period (weeks) during which stroke risk is increased. Improved contractility immediately after cardioversion may prevent arrhythmia progression. In addition, it may reduce the stroke risk. Vernakalant is a new antiarrhythmic drug able to convert atrial fibrillation to sinus rhythm and at the same time increase atrial contractility. The latter has not yet been shown in humans and is subject of the present investigation. Our hypothesis is that in humans the contractility of the atria is higher after administration of vernakalant compared to flecainide. If indeed vernakalant improves atrial contractility after cardioversion further studies into the effect on long-term arrhythmia progression and stroke prevention may follow.

ELIGIBILITY:
Inclusion Criteria:

* persistent AF or paroxysmal AF
* eligible for treatment with vernakalant or flecainide infusion to restore sinus rhythm
* receiving adequate anticoagulant therapy (or having an episode of AF lasting < 24 hours)

Exclusion Criteria:

* refusal or inability to give informed consent to participate in this study
* atrial flutter
* contra-indications for receiving vernakalant or flecainide according to MUMC+ protocol (unstable hemodynamic condition, LVEF < 40%, inadequate potassium levels, acute ischaemia, sinus node dysfunction)
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Atrial contractility measured by echocardiography | After successful cardioversion to sinus rhythm (this can be during infusion of medication or during the first hour after infusion) an echocardiography will be performed within one hour.
  Echocardiography will be performed when the patient has sinus rhythm. Transmitral flow will be measured by pulsed Doppler from an apical four chamber view. Peak velocities of the early filling (E) wave and atrial filling (A) will be determined. We will also determine the E/A ratio and the atrial volumes and the total atrial conduction time (PA-TVI).

SECONDARY OUTCOMES:
Conversion to sinus rhythm | Within one hour after drug administration
  Heart rhythm will be assessed on monitor and confirmed on ECG.
Recurrence of AF | At one month follow-up
  Heart rhythm will be assessed by ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Crijns, MD, PhD, Principal Investigator — Maastricht University Hospital
Locations (1):
- Maastricht University Hospital, Maastricht, Netherlands